CLINICAL TRIAL: NCT04481152
Title: Impact of Environmental Exposures on Tumor Risk in Subjects at Risk of Hereditary SDHx-related Paragangliomas, Pilot Phase
Brief Title: Impact of Environmental Exposures on Tumor Risk in Subjects at Risk of Hereditary SDHx Paraganglioma
Acronym: PGL-EXPO-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); ANSES (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191007; 2020-A00567-32 (Other: ANSM)
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Genetic Predisposition; SDH Gene Mutation; Environmental Exposure
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of the pilot phase of PGLEXPO will be to assess the faisability and to precise methodology of a case-control study designed for testing the impact of environmental and professional exposures on the tumoral risk in SDHx-mutation carriers

DETAILED DESCRIPTION:
The main objective of the pilot phase of PGLEXPO will be to assess the faisability and to precise methodology of a case-control study designed for testing the impact of environmental and professional exposures on the tumoral risk in SDHx-mutation carriers.

Patients will be selected from subjects with a mutation in one of the SDHx genes. The cases will have developed a tumor, while the controls will be tumor-free. Controls will be matched to the cases according to sex, age and type of gene affected. Past exposures will be sought through a telephone questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Cases: SDHx mutation carriers diagnosed for a SDHx-related tumor
2. Controls: SDHx mutation carriers with no SDHx-related tumor

Exclusion Criteria:

Incapacity to exercise free and informed consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 cases and 50 controls will be enrolled in a single referral center where they are regurlarly managed and followed for a SDHx-related tumor risk. They will be matched on their date of birth
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasability of the protocol of a national case/control study (PGL.EXPO2) | 2 years
  Successful pairing of 50 cases with 50 controls

SECONDARY OUTCOMES:
Feasibility of matching cases and controls | 2 years
  Proportion of cases for which a control could be identified
Ease of matching cases and controls | 2 years
  Mean number of controls matching for a case

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Paule GIMENEZ-ROQUEPLO, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared.
Supporting Information: Study Protocol
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.